CLINICAL TRIAL: NCT00003682
Title: Treatment of Metastatic Prostate Cancer That is Hormone-Independent: Evaluation of the Role of Chemotherapy on the Quality of Life of Patients. Phase II Study
Brief Title: Methylprednisolone With or Without Doxorubicin in Treating Patients With Metastatic Prostate Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of inclusions
Sponsor: UNICANCER (Other)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066784; FRE-FNCLCC-GETUG-02; EU-98058
Record Dates: First submitted 1999-11-01; First posted 2004-01-27 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Prostate Cancer
Keywords: stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Doxorubicin; Methylprednisolone

INTERVENTIONS:
Drug: doxorubicin hydrochloride
Drug: methylprednisolone

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to make cancer cells stop dividing so they stop growing or die. Combining chemotherapy with corticosteroids may be an effective treatment for prostate cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of methylprednisolone with or without doxorubicin in treating patients who have metastatic prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the effect of weekly doxorubicin on the quality of life of patients with metastatic, hormone-refractory, symptomatic prostate cancer. II. Determine the contribution of this treatment on control of pain in these patients. III. Determine the toxicity of this regimen in these patients. IV. Determine the objective response and biological observations in these patients after this treatment. V. Determine the effect of this regimen on survival of these patients.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to one of two treatment arms. Arm I: Patients receive methylprednisolone IV weekly for 3 months. Arm II: Patients receive methylprednisolone IV and doxorubicin IV weekly for 3 months. Quality of life is assessed before treatment, every 4 weeks during treatment, and then every 3 months. Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 160 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven, symptomatic prostate cancer Appearance or aggravation of clinical symptoms with progression of disease Bone pain OR Urethral compression OR 20% decrease in performance status Metastatic disease Local-regional or distant secondary tumors Documented radiologically or scintigraphically Hormone-refractory as defined by progression while on hormone treatment (simple castration or complete androgen blockage) Progressive disease No urethral or cervical stenosis Increase of greater than 25% prostatic volume on endorectal echography No documentation by PSA increase or imagery only Hormone castration verified by testosterone less than 0.5 ng/mL No history of CNS metastases

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: Karnofsky 60-100% Life expectancy: No specified Hematopoietic: Neutrophil count greater than 1500/mm3 Platelet count greater than 100,000/mm3 Hemoglobin greater than 9 g/dL Hepatic: Bilirubin less than 1.5 times normal Renal: Creatinine less than 1.6 mg/dL Cardiovascular: Ventricular ejection fraction at least 50% Other: No contraindication to anthracycline treatment No prior primary cancer except basal cell skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Arm I: No concurrent chemotherapy Endocrine therapy: At least 1 month since prior hormone therapy, including estramustine, except LHRH agonists, which continue Arm I: No concurrent estramustine Radiotherapy: At least 3 months since prior strontium 89 No concurrent strontium Surgery: See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 1998-10; Primary Completion 2001-03 (Actual); Study Completion 2001-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Culine, MD, Study Chair — Institut du Cancer de Montpellier - Val d'Aurelle
Locations (15):
- France (15):
  - Institut Sainte Catherine, Avignon
  - Centre de Lute Contre le Cancer,Georges-Francois Leclerc, Dijon
  - Centre Leon Berard, Lyon
  - Institut J. Paoli and I. Calmettes, Marseille
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Centre Antoine Lacassagne, Nice
  - C.H.U. - Hopital Gaston Doumergue, Nîmes
  - Institut Mutualiste Montsouris, Paris
  - Hotel Dieu de Paris, Paris
  - Institut Jean Godinot, Reims
  - Centre Eugene Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Centre Rene Huguenin, Saint-Cloud
  - Centre Hospitalier General de Saint Nazaire, Saint-Nazaire